CLINICAL TRIAL: NCT05228158
Title: A Post-marketing Observational Study of Tazemetostat on Safety in Patients With Relapsed or Refractory Follicular Lymphoma With EZH2 Gene Mutation in Japan
Brief Title: A Study of Tazemetostat on Safety in Participants With Relapsed or Refractory Follicular Lymphoma With Enhancer of Zeste Homolog 2 (EZH2) Gene Mutation in Japan
Status: Active, not recruiting | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7438-M081-501
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma, Follicular
Keywords: E7438; Tazemetostat; Tazverik
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Tazemetostat: Participants with relapsed or refractory follicular lymphoma with EZH2 gene mutation will receive Tazemetostat 800 milligram (mg), tablet, orally, twice daily or as per physicians discretion in routine clinical practice. All the participants will be observed for up to Week 52 prospectively.
  Interventions: Drug: Tazemetostat

INTERVENTIONS:
Drug: Tazemetostat — Tazemetostat oral tablets.
  Other Names: Tazverik

SUMMARY:
The primary purpose of the study is to investigate the safety of tazemetostat in participants with relapsed or refractory follicular lymphoma with EZH2 gene mutation under daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with relapsed or refractory follicular lymphoma with EZH2 gene mutation
2. Participants treated with tazemetostat

Exclusion Criteria:

1. Participants with a history of hypersensitivity to any ingredient of Tazverik

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with relapsed or refractory follicular lymphoma with EZH2 gene mutation will be enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Drug Reactions (ADRs) | Up to Week 52
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. Adverse events (AEs) with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Serious ADRs | Up to Week 52
  Serious ADRs are defined as any untoward medical occurrence or effect that at any dose resulted in death or life-threatening conditions or required hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect or medically important condition.

SECONDARY OUTCOMES:
Number of Participants With ADRs Based on Participant Background Factors | Up to Week 52
  Number of participants with ADRs such as myelosuppression and infection based on participants background factors will be reported. Participant background factors will be sex, age, height, weight, clinical stage (Ann Arbor classification), the presence or absence of B symptoms, Eastern Cooperative Oncology Group Performance Status (ECOG-PS), complications, past history and history of drug allergy.
Percentage of Participants with Overall Response | Up to Week 52
  Overall response rate is defined as a percentage of participants who achieved a best response including complete response (CR) or partial response (PR) based on Revised Response Criteria for Malignant Lymphoma (Cheson, 2007). CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.

CONTACTS AND LOCATIONS:
Locations (135):
- Japan (135):
  - Eisai Trial Site 131, Komaki-shi, Aichi-ken
  - Eisai Trial Site 199, Konan-shi, Aichi-ken
  - Eisai Trial Site 21, Nagakute-shi, Aichi-ken
  - Eisai Trial Site 106, Nagoya, Aichi-ken
  - Eisai Trial Site 156, Nagoya, Aichi-ken
  - Eisai Trial Site 174, Nagoya, Aichi-ken
  - Eisai Trial Site 91, Nagoya, Aichi-ken
  - Eisai Trial Site 170, Okazaki-shi, Aichi-ken
  - Eisai Trial Site 181, Seto-shi, Aichi-ken
  - Eisai Trial Site 130, Toyohashi, Aichi-ken
  - Eisai Trial Site 226, Toyokawa-shi, Aichi-ken
  - Eisai Trial Site 133, Toyota-shi, Aichi-ken
  - Eisai Trial Site 205, Yatomi-shi, Aichi-ken
  - Eisai Trial Site 240, Akita, Akita
  - Eisai Trial Site 234, Hirosaki-shi, Aomori
  - Eisai Trial Site 96, Hirosaki-shi, Aomori
  - Eisai Trial Site 119, Chiba, Chiba
  - Eisai Trial Site 5, Kashiwa-shi, Chiba
  - Eisai Trial Site 195, Matsudo-shi, Chiba
  - Eisai Trial Site 25, Matsuyama, Ehime
  - Eisai Trial Site 176, Fukuoka, Fukuoka
  - Eisai Trial Site 227, Fukuoka, Fukuoka
  - Eisai Trial Site 46, Fukuoka, Fukuoka
  - Eisai Trial Site 134, Iizuka-shi, Fukuoka
  - Eisai Trial Site 230, Kitakyusyu-shi, Fukuoka
  - Eisai Trial Site 252, Aizuwakayam-shi, Fukushima
  - Eisai Trial Site 82, Iwaki, Fukushima
  - Eisai Trial Site 244, Koriyama-shi, Fukushima
  - Eisai Trial Site 125, Ogaki-shi, Gifi
  - Eisai Trial Site 27, Gifu, Gifu
  - Eisai Trial Site 28, Gifu, Gifu
  - Eisai Trial Site 45, Fujioka-shi, Gunma
  - Eisai Trial Site 224, Maebashi, Gunma
  - Eisai Trial Site 235, Tatebayashi-shi, Gunma
  - Eisai Trial Site 57, Fukuyama-shi, Hiroshima
  - Eisai Trial Site 52, Hiroshima, Hiroshima
  - Eisai Trial Site 222, Asahikawa-shi, Hokkaido
  - Eisai Trial Site 198, Kitami-shi, Hokkaido
  - Eisai Trial Site 71, Kushiro, Hokkaido
  - Eisai Trial Site 167, Sapporo, Hokkaido
  - Eisai Trial Site 183, Sapporo, Hokkaido
  - Eisai Trial Site 212, Akashi-shi, Hyōgo
  - Eisai Trial Site 72, Akashi-shi, Hyōgo
  - Eisai Trial Site 31, Amagasaki-shi, Hyōgo
  - Eisai Trial Site 124, Itami-shi, Hyōgo
  - Eisai Trial Site 238, Kobe, Hyōgo
  - Eisai Trial Site 89, Kobe, Hyōgo
  - Eisai Trial Site 93, Kobe, Hyōgo
  - Eisai Trial Site 44, Nishinomiya-shi, Hyōgo
  - Eisai Trial Site 29, Hitachi-shi, Ibaraki
  - Eisai Trial Site 237, Toride-shi, Ibaraki
  - Eisai Trial Site 105, Takamatsu, Kagawa-ken
  - Eisai Trial Site 118, Kagoshima, Kagoshima-ken
  - Eisai Trial Site 207, Kanoya-shi, Kagoshima-ken
  - Eisai Trial Site 109, Ebina-shi, Kanagawa
  - Eisai Trial Site 17, Kawasaki-shi, Kanagawa
  - Eisai Trial Site 190, Kawasaki-shi, Kanagawa
  - Eisai Trial Site 87, Sagamihara-shi, Kanagawa
  - Eisai Trial Site 177, Yokohama, Kanagawa
  - Eisai Trial Site 43, Yokohama, Kanagawa
  - Eisai Trial Site 169, Yokosuka-shi, Kanagawa
  - Eisai Trial Site 9, Nankoku-shi, Kochi
  - Eisai Trial Site 253, Kumamoto, Kumamoto
  - Eisai Trial Site 55, Kumamoto, Kumamoto
  - Eisai Trial Site 26, Kyoto, Kyoto
  - Eisai Trial Site 4, Kyoto, Kyoto
  - Eisai Trial Site 56, Kyoto, Kyoto
  - Eisai Trial Site 76, Kyoto, Kyoto
  - Eisai Trial Site 122, Matsusaka-shi, Mie-ken
  - Eisai Trial Site 36, Matsusaka-shi, Mie-ken
  - Eisai Trial Site 186, Yokkaichi-shi, Mie-ken
  - Eisai Trial Site 242, Osaki-shi, Miyagi
  - Eisai Trial Site 161, Sendai, Miyagi
  - Eisai Trial Site 189, Nobeoka-shi, Miyazaki
  - Eisai Trial Site 192, Matsumoto-shi, Nagano
  - Eisai Trial Site 208, Matsumoto-shi, Nagano
  - Eisai Trial Site 127, Nagasaki, Nagasaki
  - Eisai Trial Site 251, Kashihara-shi, Nara
  - Eisai Trial Site 2, Maniwa-shi, Okayama-ken
  - Eisai Trial Site 12, Okayama, Okayama-ken
  - Eisai Trial Site 14, Okayama, Okayama-ken
  - Eisai Trial Site 178, Okayama, Okayama-ken
  - Eisai Trial Site 41, Okayama, Okayama-ken
  - Eisai Trial Site 18, Nakagami-gun, Okinawa
  - Eisai Trial Site 204, Okinawa-shi, Okinawa
  - Eisai Trial Site 164, Hirakata-shi, Osaka
  - Eisai Trial Site 49, Izumisano, Osaka
  - Eisai Trial Site 239, Kawachinagano-shi, Osaka
  - Eisai Trial Site 59, Kawachinagano-shi, Osaka
  - Eisai Trial Site 144, Osaka, Osaka
  - Eisai Trial Site 165, Osaka, Osaka
  - Eisai Trial Site 179, Osaka, Osaka
  - Eisai Trial Site 213, Osaka, Osaka
  - Eisai Trial Site 220, Osaka, Osaka
  - Eisai Trial Site 228, Osaka, Osaka
  - Eisai Trial Site 60, Osaka, Osaka
  - Eisai Trial Site 221, Sakai-shi, Osaka
  - Eisai Trial Site 233, Takatsuki-shi, Osaka
  - Eisai Trial Site 98, Toyonaka-shi, Osaka
  - Eisai Trial Site 247, Saga, Saga-ken
  - Eisai Trial Site 254, Ageo-shi, Saitama
  - Eisai Trial Site 148, Hidaka-shi, Saitama
  - Eisai Trial Site 152, Saitama-shi, Saitama
  - Eisai Trial Site 197, Saitama-shi, Saitama
  - Eisai Trial Site 140, Tokorozawa-shi, Saitama
  - Eisai Trial Site 175, Ōtsu, Shiga
  - Eisai Trial Site 223, Iwata-shi, Shizuoka
  - Eisai Trial Site 40, Izunokuni-shi, Shizuoka
  - Eisai Trial Site 88, Shizuoka, Shizuoka
  - Eisai Trial Site 201, Shimotsuke-shi, Tochigi
  - Eisai Trial Site 245, Shimotsuke-shi, Tochigi
  - Eisai Trial Site 243, Komatsushima-shi, Tokushima
  - Eisai Trial Site 101, Tokushima, Tokushima
  - Eisai Trial Site 187, Tokushima, Tokushima
  - Eisai Trial Site 158, Bunkyo-ku, Tokyo
  - Eisai Trial Site 193, Bunkyo-ku, Tokyo
  - Eisai Trial Site 225, Chiyoda-ku, Tokyo
  - Eisai Trial Site 241, Chofu-shi, Tokyo
  - Eisai Trial Site 1, Chuo-ku, Tokyo
  - Eisai Trial Site 107, Edogawa-ku, Tokyo
  - Eisai Trial Site 249, Kita-ku, Tokyo
  - Eisai Trial Site 229, Meguro-ku, Tokyo
  - Eisai Trial Site 50, Minato-ku, Tokyo
  - Eisai Trial Site 24, Shinagawa-Ku, Tokyo
  - Eisai Trial Site 162, Shinjuku-ku, Tokyo
  - Eisai Trial Site 248, Shinjuku-ku, Tokyo
  - Eisai Trial Site 159, Suginami-ku, Tokyo
  - Eisai Trial Site 231, Taito-ku, Tokyo
  - Eisai Trial Site 202, Toshima-ku, Tokyo
  - Eisai Trial Site 83, Yonago-shi, Tottori
  - Eisai Trial Site 188, Toyama, Toyama
  - Eisai Trial Site 246, Toyama, Toyama
  - Eisai Trial Site 142, Tanabe-shi, Wakayama
  - Eisai Trial Site 236, Wakayama, Wakayama
  - Eisai Trial Site 20, Sakata-shi, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.